CLINICAL TRIAL: NCT05406102
Title: Remimazolam Improves the Safety in Elderly Patients Undergoing Gastrointestinal : a Multicenter,Randomized Controlled Study
Brief Title: Remimazolam Improves the Safety in Elderly Patients Undergoing Gastrointestinal Endoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJTUIAF2020LSK-213
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2021-12

CONDITIONS: Anesthetics; Recovery; Drug Effect; Safety; Psychotropic Drugs; Anesthetics, Intravenous
Keywords: Remimazolam; Elderly; Endoscopes, Gastrointestinal; Propofol
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Patients were slowly injected of 0.08 ug/kg of sufentanil. Patients received remimazolam 0.1mg/kg to maintain sufficient sedation (sufficient sedation as judged by MOAA/S ≤ 4 for 3 consecutive measurements) during endoscopy procedure.
  Interventions: Drug: Remimazolam
- Propofol group (Active Comparator): Patients were slowly injected of 0.08 ug/kg of sufentanil for 1 min during the examination.Patients received Propofol 1.5mg/kg to maintain sufficient sedation (sufficient sedation as judged by MOAA/S ≤ 4 for 3 consecutive measurements) during endoscopy procedure.
  Interventions: Drug: Propofol group

INTERVENTIONS:
Drug: Remimazolam — Patients received an initial dose of 0.1mg/kg of remimazolam (add to 0.05 mg/kg top-ups doses to a total of up to five times within 15minutes).
  Other Names: experimental
  Arms: Remimazolam group
Drug: Propofol group — Patients received an initial dose of 1.5mg/kg of propofol(add to 0.5 mg/kg top-ups doses to a total of up to five times within 15minutes).
  Other Names: active comparator
  Arms: Propofol group

SUMMARY:
Gastroenteroscopy diagnosis and treatment drugs need to meet the needs of quick onset, quick recovery and less anesthesia complications. Remimazolam is an anesthetic sedative independently developed by China. It is a new short-acting GABA(A) receptor agonist. Remimazolam has the advantages of rapid onset, rapid recovery, antagonist, controllable degree of cardiovascular and respiratory depression, low incidence of hypotension and respiratory depression. However, elderly patients as important and special patients, there are still a lack of relevant studies and reports.

In order to verify the safety and effectiveness of remimazolam in the gastroenteroscopy treatment of elderly patients, it can reduce the incidence of intraoperative hypotension or respiratory depression rate, improve the quality of recovery of elderly patients.

DETAILED DESCRIPTION:
Patients are fasted for at least 6 hours and water for at least 2 hours. After entering the gastroscopic room, patients took 0.1 g of dacronin hydrochloride glue in the throat for about 5 minutes, instructed the patient to be in the left recumbent position and nasal catheter oxygen (4 L / min), finger oxygen and blood pressure ; after static pushing sufentanil 0.08 μg/kg, respectively, give remimazolam or propofol for sedation; MOAA/S score ≤ 3 , start gastrointestinal endoscopy, maintain MOAA/S ≤ 4 during the operation. After the end of gastrointestinal treatment, the patient is moved to the recovery room for recovery. The evaluators also assessed the incidence of blood oxygen saturation < 90%, the incidence of respiratory rate < 8 times/min, the incidence of hypotension, the time of improved aldrete≥9, the time of discharge score ≥9 points, the postoperative cognitive function, amnesia, anxiety, dizziness, pain, nausea, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60, no gender limitation;
* Patients receiving gastroscopy or gastrointestinal endoscope;
* ASA physical status score of I to III;
* 18 kg/m² < BMI < 30kg/m²;
* They clearly understand and voluntarily participate in the study and sign informed consent

Exclusion Criteria:

* Endoscopic diagnosis and treatment techniques with complex operation are required;
* Patients with respiratory management difficulties;
* Anemia or Thrombocytopenia;
* Have a history of drug abuse and/or alcohol abuse within 2 years prior to the beginning of the screening period;
* Patients with hypertension whose blood pressure is not satisfactorily controlled by antihypertensive medication (sital systolic blood pressure ≥160 mmHg at screening stage, and/or diastolic blood pressure ≥100 mmHg at screening stage);
* Allergic or contraindicated to benzodiazepines, opioids, propofol, lidocaine and their components;
* Participated in clinical trials of other drugs as a subject within the last 3 months;
* The investigator considered the patients unfit to participate in the trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-10 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hyoxemia | two hours
  The proportion of blood oxygen saturation < 90%.

SECONDARY OUTCOMES:
Incidence of respiratory depression | two hours
  The incidence of respiratory rate < 8 times/min
Incidence of hypotension | two hours
  The incidence of systolic blood pressure decreased by more than 20% before sedation or systolic blood pressure decreased to ≤ 80 mmHg.
The time of Improved Aldrete≥9 | two hours
  improved Aldrete≥9 was evaluated every 1 min after the last administration, and the time from the last administration to improved Aldrete score ≥9 .
The time of discharge score ≥9 | two hours
  the discharge score was evaluated every 3 minutes after the modified Aldrete≥9, and the time from the last administration to the discharge score ≥9.
Postoperative cognitive decline rate | two hours
  Changes in MOCA score before and after surgery
Incidence of postoperative amnesia | two hours
  incidence of anterograde and retrograde amnesia
Incidence of postoperative anxiety | two hours
  incidence of patients with generalized Anxiety Disorder Scale (GAD-7) score ≥ 10
Incidence of postoperative vertigo | two hours
  incidence of vertigo patients
Incidence of postoperative pain | two hours
  incidence of patients with visual analogue scale (VAS) ≥ 4
Adverse events | two hours
  abnormal clinical symptoms and vital signs, and abnormalities in laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (9):
- China (9):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Affiliated Tumor Hospital of Zhengzhou University, Zhengzhou, Henan
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Xian Yang Central Hospital, Xi'an, Shaanxi
  - Affiliated Hospital of Shaanxi University of traditional Chinese Medicine, Xianyang, Shaanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine, Xinjiang, Xinjiang